CLINICAL TRIAL: NCT06466694
Title: Pathways to Care-Understanding the Impact of an Indigenous Elder Co-lead in Perinatal Dialectical Behaviour Therapy (DBT) Skills Sessions in Pregnant Persons With Complex Care Needs.
Brief Title: Pathways to Care-Understanding the Impact of an Indigenous Elder Co-lead in Perinatal Dialectical Behaviour Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS26098 (H2023:234)
Record Dates: First submitted 2024-05-22; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Dialectical Behaviour Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Dialectical Behavioural Therapy (Other)
  Interventions: Behavioral: Modified Dialectical Behavioural Therapy

INTERVENTIONS:
Behavioral: Modified Dialectical Behavioural Therapy — The therapy will be co-delivered by the Elder, a perinatal psychiatrist and social worker trained in DBT. To evaluate through a patient lens content of the Dialectical Behavior Therapy (DBT) through the lens of an Indigenous Knowledge Carrier (Elder)

SUMMARY:
To integrate traditional Indigenous Knowledge with gold-standard therapy to enrich the patient experience from an anti-oppressive, culturally safe perspective for marginalized individuals with psychosocially complex pregnancies. The Knowledge Carrier does not have a prescribed way of integrating Indigenous knowledge but will respond to each patient on an individual basis depending on the needs in the current session, supporting the patients with story-telling and validation of Indigenous beliefs regarding well-being in pregnancy.

Specific Aim 1: To evaluate through a patient lens content of the Dialectical Behavior Therapy (DBT) through the lens of an Indigenous Knowledge Carrier (Elder) to make content more rich and accessible to marginalized persons.

Specific Aim 2: To provide a culturally safe space and anti-oppressive care environment for both Indigenous and non-Indigenous patients in keeping with the Truth and Reconciliation Call to Action #22

DETAILED DESCRIPTION:
Dialectical Behavior Therapy (DBT) is considered gold-standard therapy for individuals with borderline personality, and increasingly first line for addictions, coping deficits, and social instability. Participants will be asked to evaluate the integration of an Indigenous Knowledge Carrier (Elder) into a DBT program at an inner-city prenatal clinic. Patients will be pregnant or newly postpartum and qualify for DBT for routine mental health or substance associated indications. Therapy offerings will be customized to include traditional practices (ie: smudging, meditation) and teachings (ie: medicine wheel, 7 Sacred Teachings) along with standard, evidence-based content. The therapy will be co-delivered by the Elder, a perinatal psychiatrist and social worker trained in DBT. Evaluation of this modified program will be voluntary. The pre-interview guide is guided by an Appreciative Inquiry lens. The post-interview guide will be developed after analysis of the content from the pre-interview guide. Appreciative Inquiry is a qualitative research method which focuses on a strengths-based approach. The investigators will thematically analyze the data from the pre/post interviews into the predefined five stages of Appreciative Inquiry.

The investigators will utilize the Methods for Patient and Public Engagement Guide to map our research stage, level, and method of engagement. These stages include preparing for execution, data collection, data analysis, dissemination, implementation, and evaluation. Within each of these stages there are various engagement levels (consult, collaborate and partner representative) and then various methods of engagement (appreciative inquiry, discussion groups, consultations etc.) With this stepwise approach, the investigators will identify outcomes-measures that are meaningful to the population served via patient feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have their own agency and decision-making power over their health care.
* Patients may be antepartum or up to 12 weeks postpartum at the time of patient invitation.
* We will not engage minors.
* We will not engage a patient who is psychologically or physically unstable.
* We will prioritize a representative group of patients that include Black, Indigenous, People of Color (BIPOC) and represent the IPPC clinic population.

Exclusion criteria:

* Patients who are minors or who are psychologically or physically unstable.
* Our team of clinicians will screen patients prior to any initiation of engagement with these inclusion criteria as our guide, and a Pledge of Confidentiality will be obtained.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Outcomes of Modified Dialectical Therapy on marginalized pregnant patients. | 1 year
  Outcomes of Modified Dialectical Therapy with patient interviews pre and post therapy using thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Thiessen, Principal Investigator — University of Manitoba
Locations (1):
- College of Nursing, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT06466694/Prot_000.pdf